CLINICAL TRIAL: NCT01014026
Title: Human Papillomavirus DNA Testing Using Self-collected Samples for Cervical Cancer Screening: an Alternative Strategy for Unscreened Women?
Brief Title: Self-sampling and Human Papillomavirus (HPV)-Testing for Unscreened Women in Cervical Cancer Prevention
Acronym: APACHE-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: University Hospital, Tours, University Hospital, Tours
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: INCA08-KH/APACHE-1
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Uterine Cervical Neoplasms; Uterine Cervical Dysplasia
Keywords: Mass Screening; Polymerase Chain Reaction; Vaginal Smears
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia | interventions — Mass Screening

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Screening test — Two Vaginal self sampling devices and HPV test

SUMMARY:
Scientific Context

High-risk types of human papillomavirus (HPV) are the causative agents for cervical cancer. Cervical cancer screening strategies rely on periodic Papanicolaou (Pap) testing. It's well-known that this test has significantly contributed to the reduction of mortality and morbidity due to cervical cancer. In France, it now seems that the screening strategy could be optimized. The two main ways are to reach the 7 million underscreened women (mass screening, self-sampling for HPV DNA testing) and to improve the screening test (HPV DNA testing, computer-assisted cytology). Self-collected vaginal samples (SCVS) for HPV DNA testing could be a relevant screening option: this technique appears reliable and it could allow to reach women who are never or seldom screened. Currently, there is no French data on the SCVS for HPV DNA testing.

The goal of this study is to determine the performance and acceptability of a population-based strategy using self-collected vaginal samples for HPV DNA testing to reach women who are not participating in cervical cancer screening.

Description of the project

This project (APACHE-1) is a part of a project called APACHE. APACHE-1 will be dedicated to the SCVS technical validation and to the comparison between different transports medium. Nine hundred women will be recruited from the 20 to 65 years consultants in the Tours University Hospital (CHRU of Tours) and in the IRSA (health centre for routine medical checkup).

Each woman will collect 2 SCVS with a nylon flocked swab (Copan® microRheologics™). The first SCVS will be put in a vial which contains a liquid medium. The second SCVS will be put in a dry vial. Then during the speculum examination the physician will collect a cervical sample with a Rovers® Cervex-Brush™ and then rinse it into a vial containing PréservCyt ™. A blind HPV DNA testing and genotyping (Inno-LIPA HPV Genotyping ™ Extra) will be performed in the virology laboratory of the CHRU of Tours on all samples (SCVSs and cervical samples performed by a physician). The performance of the SCVS to detect cervical HPV infection will be assessed (gold standard test = HPV DNA testing on cervical samples collected by the physician).

In a second time (APACHE-2), the researchers will investigate to what extent offering home obtained SCVS leads to participation of unscreened women. APACHE-2 will be registered on Clinicaltrials as another project.

ELIGIBILITY:
Inclusion Criteria:

* Women between 20 and 65

Exclusion Criteria:

* Menstruation
* pregnant
* Inability to give informed consent
* Vaccinated against HPV 16 and 18
* Total Hysterectomy
* treatment of CIN 1, 2 or 3
* Abnormal smear in the past year
* Smear in the past 2 years
* Virgin

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 734 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Concordance between the three HPV tests | End of the study

CONTACTS AND LOCATIONS:
Overall Officials: Ken HAGUENOER, Study Director — François Rabelais University, Public Health Laboratory, Tours, France
Locations (5):
- France (5):
  - IRSA 37, La Riche
  - IRSA 72, Le Mans
  - Service d'Orthogénie, CHRU Tours, Tours
  - Service de Gynécologie, CHRU Tours, Tours
  - Association Paul Metadier, Tours